CLINICAL TRIAL: NCT04785365
Title: An Open-Label, Multi-Centre Phase II Study Evaluating the Long-Term Safety and Clinical Activity of Neoantigen Reactive T Cells in Patients Who Have Previously Received ATL001 in a Clinical Trial
Brief Title: Long-Term Follow-Up Study of Patients Receiving ATL001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The long-term follow-up of patients is being migrated to the original (parent) study protocols (Trial ID: ATX-NS-001 / NCT: NCT04032847;Trial ID: ATX-ME-001 / NCT: NCT03997474). Consequently, the ATX-LTFU-001 study is being terminated by the Sponsor.
Sponsor: Achilles Therapeutics UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ATX-LTFU-001
Record Dates: First submitted 2021-03-01; First posted 2021-03-05 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Melanoma; Advanced Non Small Cell Lung Cancer
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: ATL001 (Other): Patients who have previously received ATL001 in a clinical trial will be evaluated in this trial for long-term safety and clinical activity.
  Interventions: Other: Biological: ATL001
- Patients who have previously received ATL001 in study ATX-NS-001 or study ATX-ME-001 (Other): Patients who have previously received ATL001 in study ATX-NS-001 or study ATX-ME-001
  Interventions: Other: Biological: ATL001

INTERVENTIONS:
Other: Biological: ATL001 — No investigational product will be administered

SUMMARY:
This is an Open-Label, Multi-Centre Phase II study to evaluate the long-term safety and clinical activity of ATL001, previously administered intravenously to patients in Study ATX-NS-001 (NCT04032847) or Study ATX-ME-001 (NCT03997474).

DETAILED DESCRIPTION:
Up to 90 patients with advanced non-small cell lung cancer ( NSCLC) or metastatic or recurrent melanoma will be enrolled after either: completing 2 years of follow-up visits in study ATX-NS-001 or study ATX-ME-001; or voluntary withdrawal from these studies prior to the completion of the 2 year of follow-up period.

Each patient will be followed up for a minimum period of 5 years, or until death if sooner, in this Long-Term Follow Up Protocol.

For patients who are still alive after 5 years of follow-up, survival data will continue to be collected until the end of the study, which will occur when the last patient has completed 5 years of follow-up withdraws from study or has died.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have given written informed consent to participate in the study.
2. Patients must have received ATL001 in a previous Clinical Trial.
3. Patients must be considered, in the opinion of the Investigator, capable of complying with the protocol requirements.

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events to evaluate long-term Safety and Tolerability of ATL001 | Every 4 months to 60 months; then every 6 months until death or until the end of the study, whichever came first, assessed up to 84 months.
  Evaluate the frequency and severity of adverse events related or possibly related to ATL001
Assessment of autoimmune adverse events | Every 4 months to 60 months; then every 6 months until death or until the end of the study, whichever came first, assessed up to 84 months.
  Evaluate the frequency and severity of autoimmune adverse events
Assessment of new malignancies | Every 4 months to 60 months; then every 6 months until death or until the end of the study, whichever came first, assessed up to 84 months.
  Evaluate the frequency and severity of new malignancies
Assessment of the use of medications to manage ATL001-related toxicities | Every 4 months to 60 months; then every 6 months until death or until the end of the study, whichever came first, assessed up to 84 months.
  Evaluate the use of medications to manage ATL001-related toxicities

SECONDARY OUTCOMES:
Disease Assessment for Duration of Response ( DoR) | Maximum 60 months.
  Evaluate the endpoint of DoR as assessed by the Investigator and Independent Central Review (ICR), per RECIST v1.1
Disease Assessment for Progression Free Survival (PFS) | Maximum 60 months.
  Evaluate the endpoint of PFS as assessed by the Investigator and ICR, per RECIST v1.1
Disease Assessment for Time to First Subsequent anti-cancer Therapy (TFST) | Maximum 60 months.
  Evaluate the endpoint of TFST
Assessment for Overall Survival (OS) | 6 months until death or until the end of the study, whichever came first, assessed up to 84 months
  Evaluate the endpoint of OS by the Investigator
Assessment for cancer-related medical resources | Maximum 60 months.
  Evaluate the endpoint of cancer-related medical resourcesATL001 therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Achilles Therapeutics UK Limited
Locations (1):
- University College London Hospital (UCLH) NHS Foundation Trust, University College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ATX-NS-001 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT04032847?term=achilles+therapeutics&draw=2&rank=1
- See also: ATX-ME-001 Clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT03997474?term=achilles+therapeutics&draw=1&rank=2